CLINICAL TRIAL: NCT01381835
Title: Phase I, Open-label Trial to Investigate the Effect of Severe Renal Impairment on the Pharmacokinetics and Safety of TMC435
Brief Title: TMC435-TiDP16-C126 - Trial to Investigate the Effect of Severe Renal Impairment on the Pharmacokinetics and Safety of TMC435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017953; TMC435-TiDP16-C126 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C126; TMC435-C126; TMC435; HCV; Hepatitis C; Hep C; severe renal impairement
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental): TMC435 150 mg capsule once daily for 7 days
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — 150 mg capsule once daily for 7 days

SUMMARY:
The purpose of this study is to assess the steady-state pharmacokinetics of TMC435 in participants with severe renal impairment and to compare these with the TMC435 pharmacokinetics in matched participants with normal renal function. We will also study the short-term safety and tolerability of TMC435, when administered in participants with severe renal impairment and in participants with normal renal function. Steady-state is a term that means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body, and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is a protease inhibitor (PI) and is being investigated for treatment of chronic hepatitis C virus (HCV) infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). The result of this study may provide dosing recommendations for TMC435 in patients with severe renal impairement. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), to investigate the effect of severe renal impairment on the pharmacokinetics and safety of TMC435. Severe renal impairment will be defined by an estimated glomerular filtration rate (eGFR) = 29 mL/min/1.73m2. Participants with severe renal impairment are only allowed in this study if they are not on dialysis. Normal renal function will be considered as an eGFR = 80 mL/min/1.73m2. eGFR is a measured filtering capacity of the kidneys. The trial population will consist of a total of 16 male or female participants. Eight (8) healthy participants with a normal renal function and 8 participants with severe renal impairment will be included. A healthy participant will be matched to a participant with severe renal impairment with regards to sex, race, age (± 10 years), and body mass index (BMI) (± 20%). Dosing of the matched healthy participants can only start once the corresponding participants with severe renal impairment has completed Day 10 assessments (including physical examination). All participants will receive TMC435150 mg once a day (q.d.) for 7 days under fed conditions. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, on Day 1, Day 7, at the follow-up visit at 1 week after last dose of study medication and at the follow-up visit at 4-5 weeks after last dose of study medication. A physical examination will be performed at screening, on Day -1 (= day before first medication intake), on Day 10 and during the follow-up visits. A full pharmacokinetic profiles of bound TMC435 will be determined on Day 7 up to 72 hours postdose. In addition, unbound TMC435 plasma concentrations will be determined at specified timepoints. Safety and tolerability will be monitored throughout the trial. Participants will be admitted to the unit on Day-1 and discharged on Day10. Each participant will receive orally 150 mg TMC435, q.d. for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months before study screening. Body Mass Index of 18.0 to 35.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests, vital signs, and electrocardiogram.
* Volunteers with severe renal impairment must also meet the following inclusion criteria: 1. Consistent with the disease process causing the chronic renal failure and associated symptoms, otherwise judged to be in good health in the opinion of the investigator on the basis of a medical evaluation (including a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening). 2. Volunteers with severe renal impairment with an estimated glomerular filtration rate (eGFR) = 29 mL/min/1.73m2, who are not on dialysis and are not expected to start dialysis in the next 3 months. 3. Severity of renal disease has to be stable: no significant change in renal function as evidenced by the serum creatinine value within ±25% from the last determination, obtained within at least 6 months before study entry. 4. Volunteers with diabetes mellitus can be included provided that the disease is controlled (i.e., HbA1c <7%). 5. Stable treatment regimen for renal impairment from 2 months prior to treatment start. Diuretics are allowed when needed. 6. Concomitant medications to treat underlying disease states or medical conditions related to renal insufficiency may be used, except when specifically excluded by name or pharmacological class, and provided that dosages are stable for at least 2 months prior to treatment start.
* Matched healthy participants must also meet the following inclusion criteria: 1. Judged to be in good health in the opinion of the investigator on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, ECG, vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening. 2. Normal renal function, i.e., eGFR = 80 mL/min/1.73m2. 3. Matched to a participant with severe renal impairment with regards to sex, race, age (± 10 years) and BMI (± 20%). Exclusion Criteria:
* Infection with hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* History of or any current medical condition which could impact the safety of the participant in the study
* Having previously been dosed with TMC435 in a multiple-dose trial with TMC435
* Having previously been dosed with TMC435 in more than 3 single-dose trials with TMC435.
* Participants with severe renal impairment must also not have any of the following characteristics: 1. History of renal transplant or renal carcinoma. Participants with a history of renal carcinoma who have been cancer free for at least 5 years may be included. 2. Uncontrolled hypertension. 3. Hepatorenal syndrome. 4. Imminent renal replacement therapy (i.e., during the trial period).
* Matched healthy subjects must also not have the following characteristics: History of congenital or hereditary kidney disease (including polycystic kidney disease), nephrectomy, renal transplant or nephrolitiasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in the steady-state plasma pharmacokinetics of TMC435 following administration in participants with severe renal impairement, as compared to the matching healthy participants. | Measured on Day 5-10.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Prague, Czechia

REFERENCES:
- See also: A Phase I, open-label trial to investigate the effect of severe renal impairment on the pharmacokinetics and safety of TMC435 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1120&filename=CR017953_CSR.pdf